CLINICAL TRIAL: NCT00078260
Title: A Randomized Phase 3 Study of Two Doses of Alimta in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer Who Have Failed a Prior Platinum-Containing Chemotherapy
Brief Title: A Comparison of Two Doses of Pemetrexed in Patients Who Have Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8433; H3E-MC-JMGX (Other: Eli Lilly and Company)
Record Dates: First submitted 2004-02-20; First posted 2004-02-24 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: pemetrexed
- B (Experimental)
  Interventions: Drug: pemetrexed

INTERVENTIONS:
Drug: pemetrexed — A: 500 mg/m2, IV, q 21 days until disease progression
  B: 900 mg/m2, IV, q 21 days until disease progression

SUMMARY:
The purposes of this study are to determine:

* the safety of pemetrexed and any side effects that might be associated with it
* how much pemetrexed should be given to patients.

It is possible that information collected during this study will be analyzed by the Sponsor in the future to evaluate pemetrexed for other possible uses or for other medical or scientific purposes other than those currently proposed.

Although pemetrexed has been shown to be effective in some patients with non-small-cell lung cancer, pemetrexed might not have beneficial effects for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of locally advanced or metastatic (Stage III or IV at entry) non-small cell lung cancer (NSCLC) that is not amenable to curative therapy.
* Patients must have been previously treated with one platinum-containing chemotherapy regimen for locally advanced or metastatic disease. Patients are also eligible if they have received one platinum-based chemotherapy regimen as neoadjuvant or adjuvant chemotherapy, but must have received an additional chemotherapy regimen upon recurrence.
* No more than two prior systemic anti-cancer therapies will be allowed.
* Prior radiation therapy is allowed to less than 25% of the bone marrow. Prior radiation to the whole pelvis is not allowed. Prior radiotherapy must be completed at least 2 weeks before study enrollment, and the patient must have recovered from the acute toxic effects of the treatment prior to study enrollment.

Exclusion Criteria:

* Pregnancy.
* Breast-feeding.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Inability to interrupt aspirin, or other nonsteroidal anti-inflammatory agents for a 5-day period.
* Inability or unwillingness to take folic acid or vitamin B12 supplementation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 589 (Actual)
Dates: Start 2003-12; Primary Completion 2006-10 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Overall survival | baseline to date of death from any cause

SECONDARY OUTCOMES:
Progression free survival | baseline to measured progressive disease
Tumor response rate | baseline to measured progressive disease
Adverse events | every cycle

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Turkey (Türkiye) (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ankara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gaziantep

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Result] Cullen MH, Zatloukal P, Sorenson S, Novello S, Fischer JR, Joy AA, Zereu M, Peterson P, Visseren-Grul CM, Iscoe N. A randomized phase III trial comparing standard and high-dose pemetrexed as second-line treatment in patients with locally advanced or metastatic non-small-cell lung cancer. Ann Oncol. 2008 May;19(5):939-45. doi: 10.1093/annonc/mdm592. Epub 2008 Feb 17. PMID 18283036
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com